CLINICAL TRIAL: NCT05037396
Title: Treatment History, Demographic Characteristics, Clinical Characteristics, and Early Treatment Patterns of Patients Who Received Brolucizumab for Neovascular Age-related Macular Degeneration: IRIS Registry Study
Brief Title: Evaluation of Number of Patient Eyes That Remained on or Switched to Anti-VEGF Treatment After Initiation of Broluciumab
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CRTH258AUS12
Record Dates: First submitted 2021-07-29; First posted 2021-09-08 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Age-related Macular Degeneration (AMD)
Keywords: AMD,; brolucizumab,; anti-VEGF switchers,; treatment-naive
MeSH Terms: conditions — Macular Degeneration | interventions — brolucizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Brolucizumab: Participants received brolucizumab injection during the index period
  Interventions: Drug: Brolucizumab

INTERVENTIONS:
Drug: Brolucizumab — Participants received brolucizumab injection during the index period
  Other Names: BEOVU®

SUMMARY:
This was a retrospective cohort study to assess the treatment history, demographic characteristics, clinical characteristics, and early treatment patterns of patients who received brolucizumab for neovascular age-related macular degeneration using IRIS Registry.

DETAILED DESCRIPTION:
This was a retrospective cohort study of patients with wet AMD who received brolucizumab. Evidence was generated from the IRIS registry to describe patient treatment histories, demographic and clinical characteristics, and early treatment patterns.

Setting and study population:

IRIS Registry EHR data from 10/08/2018 to the 03/31/2020 from patients with wet AMD who initiated brolucizumab were analyzed.

Identification period of the index date: The patients fulfilling the selection criteria identified during the period from 10/08/2019 to 03/31/2020.

Index date: Defined as the date of the earliest brolucizumab injection.

Study Period: The period from 10/08/2018 to 03/31/2020.

Pre-index period: The period 12 months prior to the index date.

Post-index period: The period 4 months after the index date (not a required selection criterion; only for the assessment of select endpoints in a subgroup of patients).

ELIGIBILITY:
Inclusion Criteria:

* Patients with ≥1 brolucizumab injection
* Diagnosis of wet AMD (ICD-10: H35.3210, H35.3211, H35.3212, H35.3213, H35.3220, H35.3221, H35.3222, H35.3223, H35.3230, H35.3231, H35.3232, H35.3233, H35.3290, H35.3291, H35.3292, and H35.3293) on the index date

Exclusion Criteria:

* There were no exclusion criteria

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with wet AMD who initiated brolucizumab were analyzed in this study
Sampling Method: Non-Probability Sample
Enrollment: 9457 (Actual)
Dates: Start 2020-03-05 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Number of patients eyes with wet AMD that switched to another anti-VEGF agent (switchers) after initiation of brolucizumab within 4 months | Up to 4 months post brolucizumab injection
  To describe anti-VEGF treatment status (naive or switcher) in patients with wet AMD who initiated brolucizumab

SECONDARY OUTCOMES:
Age information | Index date
  Age information was reported
Gender information | Index date
  Gender information was reported
Number of participants: Regions | 12-month period prior to index
  Northeast, North Central, South, West, Unknown
Number of participants: Insurance type | 12-month period prior to index
  Private, Medicare, Medicare Advantage, Medicaid, Other
Number of participants: Laterality | 12-month period prior to index
  Unilateral, Bilateral
Number of participants: Race | 12-month period prior to index
  White, African American, Asian
Number of participants: Concurrent eye disease | 12-month period prior to index
  Participants were measured at the eye level for the following eye diseases: Cataracts, Posterior vitreous detachment, Epiretinal membrane, Macular hole, Vitreomacular traction, Amblyopia, Pseudophakia, Glaucoma, Diabetic macular edema, Retinal vein occlusion, Diabetic retinopathy, Myopic choroidal neovascularization
Number of participants: Provider specialty | At the brolucizumab index date defined as the date of first brolucizumab injection
  Participants were categorized based on provider specialty at date of first brolucizumab injection (e.g. Retina specialist, Ophthalmologist, etc)
Encounter location (practice location) | At the brolucizumab index date defined as the date of first brolucizumab injection
  Midwest, Northeast, South, West, Unknown
Eye location of brolucizumab injections | 12-month period prior to index
  e.g. OD [eye, right], OS [eye, left], Unspecified
Index Visual acuity (VA) | At the brolucizumab index date defined as the date of first brolucizumab injection
  Visual acuity using Snellen and approximate Early Treatment Diabetic Retinopathy Study [ETDRS] letters).
  Snellen VA ranges:
  20/12-20/20 20/25-20/40 20/50-20/160 20/200 or worse
Wet AMD diagnosis for the fellow eye | At the brolucizumab index date defined as the date of first brolucizumab injection
  Wet AMD diagnosis for the fellow eye as of the index date (Yes/No)
Visual acuity of the fellow eye | At the brolucizumab index date defined as the date of first brolucizumab injection
  Visual acuity using Snellen and approximate Early Treatment Diabetic Retinopathy Study [ETDRS] letters).
  Snellen VA ranges:
  20/12-20/20 20/25-20/40 20/50-20/160 20/200 or worse
Number of prior anti-VEGF treatments | 12-month period prior to index
  Number of anti-VEGF treatments used prior to brolucizumab at index by number of eyes were reported
Type of prior anti-VEGF treatment among switchers to brolucizumab | 12-month period prior to index
  Type of anti-VEGF agent (aflibercept, bevacizumab, ranibizumab, unlicensed bevacizumab) used immediately prior to index were reported
Prior anti-VEGF treatment sequence | 12-month period prior to index
  Prior treatment sequence(s) for previously treated eyes were reported. Continuous or Categorical (aflibercept, bevacizumab and ranibizumab)
Number of prior anti-VEGF injections received prior to brolucizumab index date | 12-month period prior to index
  Total and Per treatment prior anti-VEGF injections received prior to brolucizumab index date were reported
Injection intervals for the eyes that had received anti-VEGF injections prior to index | 12-month period prior to index
  Last injection interval, Average of last two injection intervals and Average of last three injection intervals were reported
Anti-VEGF treatment status for the fellow eye | At the brolucizumab index date defined as the date of first brolucizumab injection
  Anti-VEGF treatment endpoints for the fellow eyes with wet AMD (Naive, Switcher) were reported
Type of treatment for the fellow eye | At the brolucizumab index date defined as the date of first brolucizumab injection
  Following type of treatment for the fellow eye will be reported: aflibercept, bevacizumab, ranibizumab, brolucizumab, unlicensed bevacizumab, or none)
The number of prior anti-VEGF treatments for the fellow eye | At the brolucizumab index date defined as the date of first brolucizumab injection
  Number of prior anti-VEGF injections for the fellow eye will be reported: Continuous or Categorical (e.g. 0, 1, ≥2)
Number of brolucizumab injections received per study eye | Up to 4 months post index date
  Early treatment patterns after brolucizumab index date in anti-VEGF switcher and anti-VEGF naive patient eyes were reported
The last injection interval | Up to 4 months post index date
  The length of the interval between the final two injections was reported
The first injection interval after switch compared to last injection interval with a prior treatment | Up to 4 months post index date
  Longer, same or shorter interval were reported
Type of anti-VEGF agent initiated after switching from index brolucizumab | First 3 months after switching from index brolucizumab
  Thr type of anti-VEGF agent initiated in the first 3 months after switching from index brolucizumab. were reported

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigational site, East Hanover, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Results for CRTH258AUS12 from the Novartis Clinical Trials Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17857